CLINICAL TRIAL: NCT04359004
Title: A Study to Evaluate the Effect of Vagus Nerve Stimulation in Patients Undergoing Ventricular Tachycardia (VT) Ablation
Brief Title: A Study to Evaluate the Effect of Vagus Nerve Stimulation in Patients Undergoing VT Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kalyanam Shivkumar, MD, PhD, Director, UCLA Cardiac Arrhythmia Center & EP Programs, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-001929; OT2OD028201 (NIH)
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Arrhythmia; Ventricular Tachycardia (VT)
Keywords: Arrhythmia; Vagus Nerve Stimulation (VNS); Activation Recovery Interval (ARI)
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia, Ventricular | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Vagus Nerve Stimulation (VNS) — Vagus Nerve Stimulation (VNS) will be performed percutaneously through the internal jugular vein during the patient's routine VT ablation procedure. The nerve will be stimulated using standard pacing systems used for clinical purposes. A series of stimulation frequencies and pulse widths will be used to define optimal effects and 'dosing'. Activation recovery interval (ARI) will be measured from the unipolar electrograms. In addition, heart rate and blood pressure responses will be continuously recorded.

SUMMARY:
Vagus nerve stimulation (VNS) has been shown to be beneficial in multiple studies including heart failure. The goal of this clinical investigation is to gain additional information about how vagus nerve stimulation relates to abnormal heart rhythms. The outcomes of this study will help researchers design new therapies for patients that have complex and life-threatening ventricular arrhythmias.

DETAILED DESCRIPTION:
This study is a non-randomized, prospective study in 6 patients with scar mediated ventricular arrhythmias who are scheduled to undergo a catheter ablation procedure. The study will last up to 30 minutes in the cardiac electrophysiology lab. Cervical VNS is performed percutaneously through the internal jugular vein during the patient's routine ventricular tachycardia (VT) ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Presence of structural heart disease as defined as EF ≤ 50% or presence of ventricular scar as detected by imaging modalities or electroanatomic mapping, hypertrophic cardiomyopathy, cardiac sarcoidosis, or arrhythmogenic right ventricular cardiomyopathy.
* Age > 18 years old
* Underlying sinus rhythm with heart rate > 50 bpm.
* Provision of signed/dated informed consent and stated willingness to comply with all study procedures

Exclusion Criteria:

* Active ongoing cardiac ischemia as assessed by: ECG, cardiac enzymes, symptoms, coronary angiography with evidence of significant epicardial coronary stenosis (>70%), or stress testing. (Note: positive troponin assay due to Internal Cardiac Defibrillator (ICD) shocks is not an exclusion criterion).
* Status post orthotopic heart transplantation
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal).
* Unable or unwilling to comply with protocol requirements.
* Known channelopathy such as long QT syndrome, Brugada syndrome, and catecholaminergic polymorphic VT.
* Known peripheral neuropathy or history of autonomic dysfunction due to non-cardiac causes.
* New York Heart Association Class IV heart failure or use of current vasopressor medications
* Incessant VT
* Persistent atrial fibrillation
* Frequent premature atrial or ventricular contractions
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
The change in ventricular action potential duration during stimulation compared to baseline in msec | Up to 30 minutes or completion of the vagus nerve stimulation

SECONDARY OUTCOMES:
The change in blood pressure during stimulation compared to baseline in mmHg. | Up to 30 minutes or completion of the vagus nerve stimulation
The change in heart rate during stimulation compared to baseline in beats per minute | Up to 30 minutes or completion of the vagus nerve stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Kalyanam Shivkumar, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaseghi M, Salavatian S, Rajendran PS, Yagishita D, Woodward WR, Hamon D, Yamakawa K, Irie T, Habecker BA, Shivkumar K. Parasympathetic dysfunction and antiarrhythmic effect of vagal nerve stimulation following myocardial infarction. JCI Insight. 2017 Aug 17;2(16):e86715. doi: 10.1172/jci.insight.86715. eCollection 2017 Aug 17. PMID 28814663